CLINICAL TRIAL: NCT02511509
Title: Comparison of the Efficacy and Safety of the Bifrontal Electroconvulsive Therapy (ECT) and the Standard Bitemporal ECT in the Treatment of Patients With Schizophrenia
Brief Title: Bifrontal and Bitemporal Electroconvulsive Therapy (ECT) in Treatment of Patients With Schizophrenia
Acronym: ESBECT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Lodz (Other)
Responsible Party: Principal Investigator, Jakub Kazmierski, PhD, Medical University of Lodz
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RNN/535/10/KB
Record Dates: First submitted 2015-07-09; First posted 2015-07-30 (Estimated); Last update posted 2016-10-03 (Estimated); Status verified 2016-09

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Electroconvulsive Therapy; Bifrontal ECT; Bitemporal ECT; Cognitive functions; Postictal delirium
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bifrontal electroconvulsive therapy (Experimental): The ECT courses will be held twice or three times a week. There is no stated minimal nor maximal number of ECT courses. If there is no improvement after 12 courses, the ECT will be regarded as ineffective.
  Interventions: Device: Bifrontal electroconvulsive therapy
- Bitemporal electroconvulsive therapy (Active Comparator): The ECT courses will be held twice or three times a week. There is no stated minimal nor maximal number of ECT courses. If there is no improvement after 12 courses, the ECT will be regarded as ineffective.
  Interventions: Device: Bitemporal electroconvulsive therapy

INTERVENTIONS:
Device: Bifrontal electroconvulsive therapy — The centre of each electrode will be placed 4-5 cm above the outer canthus of the eye along a vertical line perpendicular to a line connecting the pupils.
  Arms: Bifrontal electroconvulsive therapy
Device: Bitemporal electroconvulsive therapy — The centre of the stimulus electrodes will be applied 2-3 cm above the midpoint of the line connecting the outer canthus of the eye and the external auditory meatus on each side of the individual's head.
  Arms: Bitemporal electroconvulsive therapy

SUMMARY:
Electroconvulsive therapy has been used in clinical practice since 1938, a number of randomized trials found significant differences favoring ECT in response rates between individuals with depression receiving real and sham ECT. Results of early studies performed on patients with schizophrenia weren't so clear, only few of these trials found appreciable differences between real and sham ECT in clinical outcome. The recent, more reliable studies have found that ECT is efficacious on different symptoms which might be present in the course of schizophrenia, for example, psychotic and affective ones, as well as suicidality. The serious complications of electroconvulsive therapy are rare, however, more frequent side effects may include cognitive impairment and postictal delirium. Thus, the researchers try to develop new, more effective and less harmful procedures of ECT, like bifrontal electrodes. The available studies revealed that bifrontal ECT has equal efficacy to bitemporal ECT with less cognitive impairment, but the literature examining this placement is limited to major depressive disorder and the results are inconsistent. In the worldwide literature there is lack of studies regarding the use of bifrontal ECT among patients with schizophrenia. It is interesting how bifrontal ECT would affect axial symptoms of schizophrenia, since the electrodes in this procedure are placed over the brain areas responsible for negative symptoms. This randomized, double blind study is going to assess whether the bifrontal ECT is more effective in the treatment of positive and negative symptoms of schizophrenia, has less harmful impact on the cognitive functions and decrease the frequency and severity of postictal delirium comparing to the bitemporal ECT. Moreover, as the first worldwide will assess the brain dopaminergic activity with the use of PET in the patients with schizophrenia after ECT and the impact of the ECT on the concentration of such neurotrophins as brain-derived neurotrophic factor-BDNF, neuron specific enolase-NSE and protein S100B.

ELIGIBILITY:
Inclusion Criteria:

* The patients who met Diagnostic and Statistical Manual-DSM-V criteria for schizophrenia (apart from residual type)
* The patients qualified for ECT according the standard protocol
* Antipsychotic treatment with dibenzepins according to the following scheme: the dose of clozapine not higher than 450mg, the dose of olanzapine not higher than 20mg and the dose of quetiapine not higher than 600mg per day
* If needed concomitant treatment allowed with hydroxyzine (max. 100mg per day) and lorazepam (max. 4mg per day)
* Anaesthesia conducted with the use of suxamethonium chloride, propofol and atropine

Exclusion Criteria:

* The lack of patient's consent
* Mental retardation confirmed with the psychological and psychiatric examination (IQ<70; fulfilled DSM-V criteria for mental retardation)
* Dementia diagnosed on the basis of DSM-V criteria
* Substance abuse during the year prior study enrolment or substance addiction
* The presence of symptoms which met DSM-V criteria for affective episode (an episode of mania, hypomania or depression)
* The ECT conducted during 6 months prior the study enrolment
* The history of previous ineffective ECT
* The need for antipsychotic treatment other than derivatives of dibenzothiazepines or in doses higher than 450mg of clozapine, 20mg of olanzapine and 600mg of quetiapine per day
* The women in the generative period who do not use effective contraception (sexual abstinence, contraceptives, intrauterine device, mechanical contraceptive devices)
* The need for use of other than suxamethonium chloride, propofol and atropine anaesthetics and concomitant medications

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-09; Primary Completion 2018-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Positive and Negative Syndrome Scale | up to 5 weeks
  Assessment conducted on baseline, after 6th, 12th and the last ECT.
Clinical Global Impression | up to 5 weeks
  Assessment conducted on baseline, after 6th, 12th and the last ECT.
Memorial Delirium Assessment Scale | up to 5 weeks
  Assessment conducted after the each ECT course.
Confusion Assessment Method | up to 5 weeks
  Assessment conducted after the each ECT course.
Verbal Memory Test | up to 5 weeks
  Assessment conducted on baseline, after the 6th ECT and one week after the last ECT (24 hours after each ECT course).
Visual Memory Test | up to 5 weeks
  Assessment conducted on baseline, after the 6th ECT and one week after the last ECT (24 hours after each ECT course).
Finger Tapping Test | up to 5 weeks
  Assessment conducted on baseline, after the 6th ECT and one week after the last ECT (24 hours after each ECT course)
Symbol Digit Coding Test | up to 5 weeks
  Assessment conducted on baseline, after the 6th ECT and one week after the last ECT (24 hours after each ECT course)
Stroop Test | up to 5 weeks
  Assessment conducted on baseline, after the 6th ECT and one week after the last ECT (24 hours after each ECT course)
Shifting Attention Test | up to 5 weeks
  Assessment conducted on baseline, after the 6th ECT and one week after the last ECT (24 hours after each ECT course)
Continuous Performance Test | up to 5 weeks
  Assessment conducted on baseline, after the 6th ECT and one week after the last ECT (24 hours after each ECT course).

SECONDARY OUTCOMES:
Positron Emission Tomography to assess the impact of ECT on the dopaminergic system activity | up to 5 weeks
  Assessment conducted before the first and after the last ECT course.
The concentration of brain-derived neurotrophic factor. | up to 5 weeks
  The blood samples will be collected on baseline, 2 and 6 hours after the first ECT course, 2 hours after the 3rd, 6th, 9th and the last ECT course
The concentration of neuron specific enolase. | up to 5 weeks
  The blood samples will be collected on baseline, 2 and 6 hours after the first ECT course, 2 hours after the 3rd, 6th, 9th and the last ECT course
The concentration of protein S100B | up to 5 weeks
  The blood samples will be collected on baseline, 2 and 6 hours after the first ECT course, 2 hours after the 3rd, 6th, 9th and the last ECT course

CONTACTS AND LOCATIONS:
Overall Officials: Iwona Kloszewska, Prof., Principal Investigator — Medical University of Lodz, Poland
Locations (1):
- Department of Old Age Psychiatry and Psychotic Disorders Medical University of Lodz, Lodz, Poland